CLINICAL TRIAL: NCT06885853
Title: Evaluation of Long-term Immunogenicity of a Boost Dose of MVA-BN Vaccine
Acronym: M-BOOST-FR
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP250053; IDRCB:2025-A00095-44 (Other: ANSM)
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Monkeypox
Keywords: Monkeypox; MVA-BN booster vaccine; HIV pre-exposure prophylaxis
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is to evaluate the long-term immunogenicity of a boost dose of MVA-BN vaccine

DETAILED DESCRIPTION:
Mpox is an endemic zoonosis in Africa, caused by the MPXV virus of which there are two clades: I (former Congo Basin) and II (former West Africa). Since 2022, clade II has emerged globally via sexual transmission, primarily among men who have sex with men (MSM), resulting in a declaration of public health emergency (PHEIC) by the WHO.

In 2023, a clade I epidemic emerged in East Africa with a high case fatality rate (3-5%). In August 2024, the WHO again declared a PHEIC after the spread of clade I to African countries with no previously reported cases and outside Africa, raising fears of higher mortality and transmission.

A 3rd generation vaccine, MVA-BN (Imvanex® /Jynneos®), initially developed against smallpox, was approved in 2022 to prevent mpox. In France, the HAS recommends post- and pre-exposure vaccination for populations at risk: MSM, trans people with multiple partners, sex workers and certain professionals. For people born before 1980 (history of smallpox vaccination), a single dose is recommended as primary vaccination, while immunocompromised subjects require 3 doses.

Data show vaccine effectiveness of 20-80% in post-exposure prophylaxis (PEP) and ~80% in pre-exposure but neutralizing antibodies become undetectable after one year. Since the summer of 2024, the HAS has recommended a booster dose 2 years after the primary vaccination, on the basis of immunogenicity studies showing an increase in seroconversion to 98.7% one month after administration, but underlines the need to have other data, in particular on the durability of this response.

A study is proposed in MSM on HIV PrEP (pre-exposure prophylaxis), a priority population for structured medical monitoring, to evaluate the immunogenicity and safety of the MVA-BN booster in this context.

ELIGIBILITY:
Inclusion Criteria:

* Men aged over 18 years
* Have received two doses of MVA-BN vaccine as an initial schedule
* Eligible for a booster dose of MVA-BN (according to the HAS recommendation)
* Be eligible and wish to initiate PrEP-HIV treatment or be followed for PrEP-HIV treatment
* Covered by social security (excluding AME)

Exclusion Criteria:

* History of mpox (virologically confirmed)
* Be under guardianship or curatorship
* Be subject to a judicial protection measure
* Have a contraindication to vaccination against mpox

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of Men who have Sex with Men (MSM), taking HIV pre-exposure prophylaxis (HIV PrEP), eligible for MVA-BN vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity a of a booster dose of MVA-BN vaccine | 12 months
  To evaluate the immunogenicity at 12 months of a booster dose of MVA-BN vaccine administered subcutaneously in HIV PrEP users.

SECONDARY OUTCOMES:
Persistence of humoral immunogenicity | 24 months
  Evaluate the persistence of humoral immunogenicity at 24 months of a booster dose, depending on the number of doses and the interval between doses
Kinetics of the humoral response | 24 months
  Study the kinetics of the humoral response as a function of the number of doses and the interval between doses
Description of cases of Mpox infection | 24 months
  Describe cases of Mpox infection based on number of doses and dose interval up to 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Liem Binh Luong Nguyen, Degree medical doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CIC 1417Cochin-Pasteur, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No